CLINICAL TRIAL: NCT01419509
Title: DNA Methylation-based Assays for Detecting Disease Spread in Rhabdomyosarcoma
Brief Title: DNA Tests in Detecting Disseminated Disease in Tumor, Blood, and Bone Marrow Samples From Patients With Rhabdomyosarcoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARST11B1; COG-ARST11B1 (Other: Children's Oncology Group); ARST11B1 (Other: Children's Oncology Group); NCI-2011-02985 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Sarcoma
Keywords: alveolar childhood rhabdomyosarcoma; embryonal childhood rhabdomyosarcoma; embryonal-botryoid childhood rhabdomyosarcoma; mixed childhood rhabdomyosarcoma; pleomorphic childhood rhabdomyosarcoma; previously untreated childhood rhabdomyosarcoma; nonmetastatic childhood soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — DNA Methylation; Microarray Analysis; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor, Blood, and Bone Marrow Samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: microarray analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: DNA analysis of tumor, blood, and bone marrow may help doctors predict if the disease has been disseminated.

PURPOSE: This research trial studies DNA tests in detecting disseminated disease in tumor, blood, and bone marrow samples from patients with rhabdomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To establish a panel of hypermethylation assays for minimal disseminated disease analysis in rhabdomyosarcoma (RMS).
* To apply the hypermethylation assays to a series of bone marrow specimens from RMS patients.

OUTLINE: Archived tumor, bone marrow, and peripheral blood samples are analyzed for DNA hypermethylation by PCR-based assays and microarray assays. Results are then compared with each patient's clinical and pathological characteristics, and outcomes. Patterns of locus hypermethylation in tumor and paired bone marrow samples are also compared.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with rhabdomyosarcoma (RMS)
* Tumor, bone marrow, and peripheral blood samples from the Children's Oncology Group D9803 trial of intermediate-risk RMS

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosed with rhabdomyosarcoma
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Panel of hypermethylation assays for minimal disseminated RMS
Detection of RMS cells in bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R. Master, MD, Principal Investigator — University of Pennsylvania